CLINICAL TRIAL: NCT01859286
Title: Improving Transfer of Care Accuracy and Information Delivery in the Emergency Department
Brief Title: Improving Signout Accuracy and Information Delivery in the Emergency Department
Acronym: SAID-ED
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Justin Mazzillo, Chief Resident - Emergency Medicine, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-11-0655
Record Dates: First submitted 2013-04-27; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Medical Errors Related to Emergency Department Sign Out

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- regular sign out process
  Interventions: Other: standardized sign out process

INTERVENTIONS:
Other: standardized sign out process — The intervention phase included was the introduction of a standardized TOC (transfer of care) process, which occurred during April and May of 2012. TOC was done at a predefined location in each section of the emergency department (Medicine and Trauma). All participating residents were given a diagram detailing the central location and seating arrangement. The outgoing attending was designated to handle all distractions or disturbances that occurred during sign out. The most senior resident coming on to shift was designated the data resident. The data resident's role was to operate a centralized computer with the ED tracking board and EMR and review pending orders, vital signs and resulted labs and radiology reports after each patient was signed out. A brief pause was implemented to allow the oncoming team to ask any questions regarding that patient's care or course. The post TOC data form and protocol were identical to that of the control phase.

SUMMARY:
The investigators sought to determine if implementing a standardized sign out process would reduce the amount of medical errors related to patient sign out. The standardized process included the following interventions: implementation of a data resident to review patients lab values, vital signs, radiologist results, and orders in real time, conducting sign out in a standardized location and using the attending physician as an "interruption manager." The investigators defined medical errors related to sign out as any piece of information was incorrectly reported or omitted during sign out that caused a change in treatment or disposition discussed during sign out. The investigators hypothesis was that implementing a standardized sign out process would lead to a decrease in the amount of sign out related errors.

ELIGIBILITY:
Inclusion Criteria:

* ED transfers of care occurring at 0700 or 1900.

Exclusion Criteria:

* Attending only handovers (1500, 2300)
* Handovers including midlevel providers (Thursday 0700, 1300).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ED Physicians. We looked at the amount of errors due to signout that ED Physicians commit with standard signout procedure and then with a revised signed out process
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Sign out related errors | 4 months

SECONDARY OUTCOMES:
perception of sign out | 1 year after implementation of revised sign out process

CONTACTS AND LOCATIONS:
Overall Officials: Nnaemeka G Okafor, MD, Principal Investigator — UT Houston Health Sciences Center at Houston Department of Emergency Medicine
Locations (1):
- Memorial Hermann Hospital - Texas Medical Center, Houston, Texas, United States